CLINICAL TRIAL: NCT00399672
Title: Evaluation of a Multi-disciplinary Approach for the Treatment of Hepatitis C in IDUs (HI-LO Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C06-0192
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C Virus Infection
Keywords: HCV; injection drug users; ribavirin; pegylated interferon; illicit drug users
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): The 4 participating sites are designated either High Intensity or Low Intensity. High Intensity sites have access to: full time specialist physicians, access to full time nurses and counselors. All weekly pegylated interferon injections will be administered by clinic staff and ribavirin will be dispensed in weekly medication pack.
  Interventions: Drug: Interferon injections and ribavirin
- 2 (Active Comparator): The 4 participating sites are designated either High Intensity or Low Intensity. In the Low intensity group, all patients will have access to: full time primary care physicians, specialist physicians and access to part time nurse or counselor by appointment. Patients will be offered the option of self or nurse administered pegylated interferon injections on an appointment basis. Ribavirin will be dispensed biweekly. The treatment medication cannot be stored at the clinic; it must be the subjects responsibility.
  Interventions: Drug: Interferon injections and ribavirin

INTERVENTIONS:
Drug: Interferon injections and ribavirin — Weekly pegylated interferon injections will be administered by clinic staff and ribavirin will be dispensed in weekly medication pack.
  Arms: 1
Drug: Interferon injections and ribavirin — Patients will be offered the option of self or nurse administered pegylated interferon injections on an appointment basis. Ribavirin will be dispensed biweekly. The treatment medication cannot be stored at the clinic; it must be the subjects responsibility.
  Arms: 2

SUMMARY:
Although injection drug users (IDUs) account for over 70% of new cases of HCV infection/year, there is no consensus on how to approach their medical care. In some Canadian centres, patients must be free of recreational drug use for as long as 6 months before being considered for HCV therapy. This is not consistent with current North American guidelines. Over the past 5 years, we have developed a successful program for the treatment of HIV infection in this population, based on a multi-disciplinary comprehensive program including directly observed therapy (DOT). Even though the duration of therapy for HCV is shorter than for HIV (as little as 6 months vs. life-long), we must address issues of administration of a weekly injection (interferon), twice daily pills (ribavirin) and the risk of significant side effects (including anxiety and depression) to successfully expand our program to treat this disease. Further, it may be that even if the program is successful, its benefits will be negated by HCV re-infection due to continued risk behaviors for its transmission.

DETAILED DESCRIPTION:
We will determine the HCV infection status of potential study subjects within a cohort of 2,000 IDUs receiving care in our centres (Appendix 1). For those who carry HCV antibodies (expected n = 1800), a test for HCV viremia and genotype will be performed. By these evaluations, we expect up to 600 individuals to be viremic and carry HCV genotype 2 or 3. Within this group, 200 consecutive patients (100/study strategy) will receive therapy for HCV, based on their eligibility to do so according to Provincial guidelines for the reimbursement of medications. Patient allocation will be according to the study site where they regularly receive care. At two sites, patients will be enrolled in a DOT program with on-site full-time nursing and counseling support (high intensity, 50 patients/site). At the other two sites, patients will receive medication on a weekly basis and will have access to part-time nursing and counseling support (low intensity, 50 patients/site). Medical follow-up will be according to current clinical standards, and the primary endpoint of the study will be the rate of sustained virologic response (SVR) six months after completion of treatment. Within the study described above, we will use standardized methodologies to calculate the total health care costs related to the treatment of HCV infection. We will also assess the effect of treatment on the quality of life (QoL) of study participants.

ELIGIBILITY:
Inclusion Criteria:

* Age > 19 years;
* Serum HCV-RNA pos;
* HCV genotype 2 or 3;
* HBsAg neg;
* serum ALT > 1.5x upper limit normal > 3 months;
* Illicit drug use in the past year;
* Agreement from each participant of childbearing age to practice contraception;
* Absence of other contraindications to the initiation of therapy as determined by the health care team;
* Ability to provide informed consent.

Exclusion Criteria:

* Any cause for chronic liver disease other than HCV (including alcohol use >350 g/wk);
* Pregnant or breastfeeding women;
* Active HBV infection;
* Hemolytic anemia;
* Decompensated cirrhosis or portal hypertension or PT-INR > 1.3 or Child-Hugh class > A;
* Active suicidal ideation, psychosis, mania or hypomania;
* Serum creatinine > 180 µg/mL;
* Hemoglobin < 120 g/L in men or 110 g/L in women;
* Platelets < 90 x 109/L;
* Neutrophils < 1.5 x 109/L;
* Active autoimmune disease;
* NYHA disease > grade 2;
* Psoriasis requiring systemic therapy;
* Active malignancy apart from non melanoma skin cancer;
* Use of systemic immunosuppressant agents;
* Prior treatment of HCV with interferon or ribavirin;
* HIV positive with CD4 count <300 cells/mm3 or receiving didanosine (due to interaction with ribavirin);
* Life expectancy < 2 years.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2007-06; Primary Completion 2010-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Rate of sustained virologic response (SVR) six months after completion of treatment.

SECONDARY OUTCOMES:
Adherence to therapy
Cost
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Brian Conway, MD, Principal Investigator — University of British Columbia
Locations (1):
- Pender Community Health Centre, Vancouver, British Columbia, Canada